CLINICAL TRIAL: NCT02287727
Title: (Bayer Study ONC-2013-036) A Phase II Single-Arm Study of Regorafenib Maintenance Therapy in Patients With T3, T4 or Node-Positive Rectal Cancer Patients Who Completed Curative-Intent Treatment
Brief Title: Regorafenib in Reducing Recurrence in Patients With Non-metastatic Rectal Cancer Who Have Completed Curative-Intent Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 246813; NCI-2014-02202 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ONC-2013-036; BAY ONC-3012-036; I 246813 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Rectal Adenocarcinoma; Stage IIA Rectal Cancer; Stage IIB Rectal Cancer; Stage IIC Rectal Cancer; Stage IIIA Rectal Cancer; Stage IIIB Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (regorafenib) (Experimental): Patients receive regorafenib PO QD on days 1-21. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Regorafenib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; Stivarga

SUMMARY:
This phase II trial studies how well regorafenib works in reducing the return of disease in patients with rectal cancer that has not spread to another place in the body who have completed curative-intent treatment. Regorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Regorafenib may also help keep cancer from coming back after it has disappeared following the initial therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 3-year disease free survival in patients with T3, T4 or node-positive rectal adenocarcinoma who received regorafenib maintenance therapy following the completion of curative-intent standard treatment.

SECONDARY OBJECTIVES:

I. To determine the cumulative incidence of local recurrence, distant recurrence and overall survival at 3 years.

II. To explore for biomarkers associated with anti-cancer effects of regorafenib maintenance therapy in curatively treated rectal cancer patients by analyzing tumor and blood samples.

OUTLINE:

Patients receive regorafenib orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 4 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the rectum that was clinically staged T3, T4 or node-positive (defined as >= N1 per American Joint Committee on Cancer [AJCC] 7th edition) that was treated with the following treatment with curative intent:

  * Curative surgical resection
  * Pre- or post-operative chemoradiation; and at least 3 months of adjuvant systemic chemotherapy (equivalent to 6 cycles of leucovorin calcium, fluorouracil, and oxaliplatin [FOLFOX] or infusional fluorouracil [5FU])
* No evidence of cancer within 28 days prior to start of study treatment; this should be determined by imaging of the chest, abdomen and pelvis by computed tomography (CT) and/or magnetic resonance imaging (MRI); staging of the chest using chest x-ray in lieu of CT and/or MRI should not be used for this purpose
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Consent to allowing his/her archival tumor tissues to be requested and analyzed; however, the non-availability or inadequate amount samples for analysis will not exclude the patient
* Platelet count >= 100,000/mm^3; blood transfusion to meet the inclusion criteria will not be allowed
* Hemoglobin (Hb) >= 9 g/dL; blood transfusion to meet the inclusion criteria will not be allowed
* Absolute neutrophil count (ANC) 1500/mm^3; blood transfusion to meet the inclusion criteria will not be allowed
* Total bilirubin =< 1.5 x the upper limits of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) =< 2.5 x ULN
* Alkaline phosphatase limit =< 2.5 x ULN
* Lipase =< 1.5 x the ULN
* Serum creatinine =< 1.5 times the ULN
* International normalized ratio (INR) of prothrombin time (PT; PT-INR) and activated partial thromboplastin time (aPTT) =< 1.5: subjects who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists per medical history; close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug; post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test
* Patients of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and, until at least 3 months after the last dose of the study drug; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patient is willing and able to take oral medications and to comply with scheduled visits, treatment plan, and study related procedures

Exclusion Criteria:

* Evidence of recurrence of rectal cancer prior to the start of study treatment
* Any previously untreated or concurrent cancer that is distinct in primary site or histology from rectal cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor; subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before starting study drug are allowed; all cancer treatments must be completed at least 3 years prior to study entry (i.e., signature date of the informed consent form)
* Anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) within 4 weeks prior to entering the study (signing of consent form) or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; patients on hormonal or bisphosphonate treatment for non-cancer related conditions are eligible
* Inability to start study treatment within 12 weeks following the completion of curative intent therapy for rectal adenocarcinoma
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication; minor procedures such as diagnostic laparoscopy, percutaneous biopsy and paracentesis within 14 days before start of study medication
* Patients who have not recovered from the surgical resection of rectal cancer such as wound dehiscence, non-healing wound, wound infection and fistula
* Prior use of regorafenib
* Gastrointestinal conditions that may significantly affect the absorption of regorafenib
* Uncontrolled hypertension (systolic pressure > 140 mmHg or diastolic pressure > 90 mmHg on repeated measurement) despite optimal medical management
* Evidence or history of bleeding diathesis or coagulopathy
* Any hemorrhage or bleeding event >= Common Terminology Criteria for Adverse Events (CTCAE) grade 3 within 4 weeks prior to start of study medication
* Have had arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 3 months prior to the initiation of study treatment
* Patients with phaeochromocytoma
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy
* Ongoing infection > CTCAE grade 2
* Patients with seizure disorder requiring medication
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Pleural effusion or ascites that causes respiratory compromise (>= grade 2 dyspnea CTCAE)
* History of organ allograft (including corneal transplant)
* Pregnant or nursing female patients
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina pectoris (defined as anginal symptoms at rest, new-onset angina within 3 months before study treatment initiation, or myocardial infarction within 6 months before study treatment initiation), cardiac arrhythmia (which require anti-arrhythmic therapy other than beta blockers or digoxin), active coronary artery disease, or psychiatric illness/social situations that would limit compliance with study requirements
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs
* Therapeutic anticoagulation with vitamin-K antagonists (e.g., warfarin) or with heparins and heparinoids; however, prophylactic anticoagulation as described below is allowed:

  * Low dose warfarin (1 mg orally, once daily) with PT-INR =< 1.5 is permitted; infrequent bleeding or elevations in PT-INR have been reported in some subjects taking warfarin while on regorafenib therapy; therefore, subjects taking concomitant warfarin should be monitored regularly for changes in PT, PT-INR or clinical bleeding episodes
  * Low dose aspirin (=< 100 mg daily)
  * Prophylactic doses of heparin
* Are taking strong cytochrome P (cytochrome P450, family 3, subfamily A, polypeptide 4 [CYP3A4]) inhibitors (e.g., clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (e.g., carbamazepine, phenobarbital, phenytoin, rifampin, St. John's wort/Hypericum perforatum)
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive study drug
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 3 years
  The DFS will be summarized using the standard Kaplan-Meier methods. The 3-year DFS rate will be estimated by a 95% confidence interval, obtained using the method proposed by Breslow and Day, using the intent-to-treat approach.

SECONDARY OUTCOMES:
Biomarkers associated with anti-cancer effects of regorafenib maintenance therapy | Up to 5 years
  The potential association between selected biomarkers and time-to-event outcomes will be evaluated using Cox regression models. Hazard ratios and corresponding confidence intervals will be obtained. All secondary analysis will be conducted at a significance level of 0.05 and, as these are more exploratory in nature, no adjustments will be made for multiple testing.
Distant recurrence | 3 years
  The potential association between selected biomarkers and time-to-event outcomes will be evaluated using Cox regression models. Hazard ratios and corresponding confidence intervals will be obtained. All secondary analysis will be conducted at a significance level of 0.05 and, as these are more exploratory in nature, no adjustments will be made for multiple testing.
Frequency of toxicity, graded according to National Cancer Institute CTCAE version 4.0 | Up to 30 days following last dose of study drug
  The frequency of toxicities will be tabulated by grade across all dose levels and cycles.
Local recurrence | 3 years
  The potential association between selected biomarkers and time-to-event outcomes will be evaluated using Cox regression models. Hazard ratios and corresponding confidence intervals will be obtained. All secondary analysis will be conducted at a significance level of 0.05 and, as these are more exploratory in nature, no adjustments will be made for multiple testing.
Overall survival | 3 years
  The potential association between selected biomarkers and time-to-event outcomes will be evaluated using Cox regression models. Hazard ratios and corresponding confidence intervals will be obtained. All secondary analysis will be conducted at a significance level of 0.05 and, as these are more exploratory in nature, no adjustments will be made for multiple testing.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Boland, Principal Investigator — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester Medical Center - Wilmont Cancer Institute, Rocherster, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio